CLINICAL TRIAL: NCT07399431
Title: Effectiveness of Theta Burst Stimulation in the Management of Methamphetamine Use Disorder in Indonesia: A Randomized Controlled Trial as a National Model for Comprehensive Management
Brief Title: Theta Burst Stimulation in the Management of Methamphetamine Use Disorder in Indonesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Kristiana Siste, Dr. dr. Kristiana Siste, Sp.KJ(K) - Head of Department of Psychiatry, Cipto Mangunkusumo General Hospital, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KET-741-2025
Record Dates: First submitted 2026-01-27; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Methamphetamine Use Disorder; Theta Burst Stimulation; Transcranial Magnetic Stimulation
Keywords: Methamphetamine Use Disorder; Theta Burst Stimulation; Cognitive Behavioral Therapy; Transcranial Magnetic Stimulation
MeSH Terms: interventions — Transcranial Magnetic Stimulation; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TBS and CBT (Experimental): During 12 days of intervention, the participants underwent 10 sessions of TBS and 12 sessions for CBT.
  Interventions: Device: Theta Burst Stimulation; Behavioral: Cognitive Behavioral Therapy
- Sham and CBT (Sham Comparator): During 12 days of intervention, the participants underwent 10 sessions of sham TBS and 12 sessions of CBT.
  Interventions: Device: Theta Burst Stimulation; Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Device: Theta Burst Stimulation — A randomized controlled trial (RCT) of 20 participants underwent TBS and CBT intervention for MUD.
  Other Names: TBS; Transcranial Magnetic Stimulation; TMS
Behavioral: Cognitive Behavioral Therapy — The cognitive behavioral therapy (CBT) for methamphetamine use disorder (MUD) was conducted in 12 sessions (1 session per day). We utilized the module adapted from the Indonesia Drug Addiction and Relapse Prevention Program (Indo-DARPP) for MUD. The CBT was delivered by trained psychiatrist in group CBT setting.
  Other Names: CBT

SUMMARY:
Methamphetamine use disorder (MUD) remains a major public health concern in Indonesia, with limited effective treatment options and high relapse rates. Theta Burst Stimulation (TBS) has emerged as a promising adjunctive intervention for reducing craving and improving clinical outcomes. This trial aims to evaluate the efficacy and safety of TBS for MUD. A RCT of 20 subjects was conducted to evalute the efficacy and safety of TBS as an adjunctive treatment to CBT in managing MUD.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18-59 years old
* Subjects diagnosed with methamphetamine use disorder without having undergone treatment, whether psychotherapy and/or psychopharmacological modalities
* Subjects are able to read and write

Exclusion Criteria:

* Subjects with severe thought process disorders, impaired perception, restless condition, severe neurological disorders, history of neuromodulation,
* Subjects refused to participate in the study
* Subjects who are pregnant
* Subjects who have radioactive implants

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2025-10-19 (Actual); Primary Completion 2025-11-03 (Actual); Study Completion 2025-11-05 (Actual)

PRIMARY OUTCOMES:
Improvement in craving for methamphetamine | Baseline (T1), day 3 (T2), day 5 (T3), day 8 (T4), and day 10 (T5)
  Cue-induced craving was measured with Visual Analog Scale (VAS) where the patient told to indicate their point of craving in a 100 mm line. The scale ranged from 0 to 10, with higher scores indicated higher craving.
Improvement in craving (tonic) for methamphetamine | Baseline (T1), day 3 (T2), day 5 (T3), day 8 (T4), and day 10 (T5)
  Tonic or baseline craving was measured using the Questionnaire for Smoking Urges modified for Methamphetamine (QSU-M) in Indonesian version. The questions were self-filled by the participants to identify their level of craving. The QSU-M is a 7-point Likert Scale (1 was strongly disagree and 7 was strongly agree) with the higher total scores indicating higher tonic craving. The total minimum score was 10 while the maximum score was 70.
Improvement in clinical severity | Baseline (T1), day 3 (T2), day 5 (T3), day 8 (T4), and day 10 (T5)
  The clinical severity was measured using the Clinical Global Impression - Severity by the psychiatrist based on the patient's condition during the day of examination. CGI is a clinician-rated instrument used to assess the patient's condition based on clinical judgment. CGI mainly rates the severity of illness assessed using a 7-point Likert scale, ranges from 1 (normal) to 7 (among the most extremely ill). Higher score indicated higher severity of addiction-related illness.

SECONDARY OUTCOMES:
Improvement in Addiction Severity | Baseline (T1) and Post-Intervention Day 12 (T6)
  Addiction Severity Index (ASI) assessed the severity of a person's addiction, through multiple domains; medical, occupational, alcohol usage, substance use, law, family/social and mental status domains. The analysis utilized composite scores of relevant questions. Higher scores indicated higher severity. The minimum composite score for each domain was 0 while the maximum score was 1.
Improvement in Depressive Symptoms | Baseline (T1) and Post-Intervention Day 12 (T6)
  The Patient Health Questionnaire-9 (PHQ-9) assessed the severity of depressive symptoms, with higher scores indicating higher severity. PHQ-9 is a 9 item with 3-point Likert scale with 0 indicates no presence of symptoms and indicates higher frequency of depression symptoms (nearly every day). The higher total scores indicates higher severity of depression, with the minimum total score of 0 and the maximum score of 27.
Improvement in Motivation to Change | Baseline (T1) and Post-Intervention Day 12 (T6)
  University of Rhode Island Change Assessment (URICA) assessed a person's readiness for change, with scores divided into four subscales: pre-contemplation, contemplation, action and maintenance. URICA is a five-point Likert scale consisting of 32 questions, ranges from 1 (strongly disagree) to 5 (strongly agree). The minimum averaged score per subscale was 1 while the maximum score was 5. The calculation was done with the formula as follow: (averaged contemplation + averaged action + averaged maintenance)/averaged pre-contemplation.
  Higher overall score indicated higher stage of change.
Improvement in Impulsivity | Baseline (T1) and Post-Intervention Day 12 (T6)
  The Barratt Impulsiveness Scale version 11 (BIS-11) assesed impulsive attitudes and behaviors. BIS-11 was a four-point Likert scales of 30 items, ranged from 1 (never/very rarely), 2 (rarely), 3 (often), and 4 (almost always). The total scores ranged from 30 to 120. Higher scores indicate higher overall impulsivity.
Improvement in Sleep Quality | Baseline (T1) and Post-Intervention Day 12 (T6)
  The Pittsburgh Sleep Quality Index (PSQI) assessed sleep quality, measuring subjective sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbances, use of sleep medications, and daytime dysfunction. PSQI consisted of different segments of questions from sleep duration, habitual efficiency, and symptoms of sleeping problems. The symptoms were measured in 4-point Likert scale where 0 indicated no difficulty and 3 indicated high difficulty of sleeping. This instrument consisted of 19 questions, yielding a global score from 0 to 21. A higher total score indicated poor sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitas Indonesia, Jakarta Pusat, Jakarta Special Capital Region, Indonesia